CLINICAL TRIAL: NCT04686396
Title: Demineralized Bone Matrix Rotator Cuff Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Arthrex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: US-1300
Record Dates: First submitted 2020-12-23; First posted 2020-12-28 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2020-12

CONDITIONS: Rotator Cuff Injuries
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to have either the addition of demineralized bone matrix to their procedure (Interpositional Group), or standard Rotator Cuff repair without demineralized bone matrix administered (Control group).
Who Masked: Participant
Masking Description: Randomization shall be performed during surgery after intra-operative inclusion/exclusion eligibility has been met.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Interpositional Group (Experimental): Demineralized bone matrix
  Interventions: Device: Demineralized bone matrix
- Control (No Intervention): Without demineralized bone matrix

INTERVENTIONS:
Device: Demineralized bone matrix — Demineralized bone matrix
  Arms: Interpositional Group

SUMMARY:
Patients undergoing rotator cuff repair surgery will experience improved tendon healing with the use of demineralized bone matrix augmentation.

DETAILED DESCRIPTION:
This is a prospective randomized study comparing the outcomes of patient undergoing rotator cuff repair with either an interpositional procedure administering demineralized bone matrix (DBM), or a control group without demineralized bone matrix. Patient outcomes will be collected and compared between the two cohorts up to a five (5) year post-operative period and will include a range of subjective and functional outcomes, along with radiographic imaging.

ELIGIBILITY:
Inclusion Criteria:

* The Subject is between the ages of 40 and 75 years.
* Subject is planning to undergo arthroscopic surgery for full thickness rotator cuff tears (RCT) of supraspinatus and infraspinatus muscles, who are candidates for demineralized bone matrix with BMC.
* Two tendon tear or tear size equal to or greater than 3cm
* Amenable to double-row repair
* Primary rotator cuff tears with or without superior labral tear and/or biceps tear)

Exclusion Criteria:

* The Subject is unable or unwilling to sign the Patient Informed Consent, approved by the Institutional Review Board.
* The Subject objects to use of allograft
* Irreparable Rotator Cuff Tear
* Complete full thickness subscapularis tears of > than the superior 1/3 of the tendon (Lafosse grade 3 and above)
* < 2 mm joint space of the glenohumeral joint on either an anteroposterior or axillary radiograph
* Recurrent shoulder instability
* Intra-articular injections (steroids) within 1 month of surgery
* RCR revisions
* Subject MRI taken more than 12 months prior to surgery
* Pregnant or planning to become pregnant during the study period
* Workman's compensation case

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
MRI | 24 weeks
  Rate of healing of the rotator cuff repair

SECONDARY OUTCOMES:
American Shoulder and Elbow Surgeons Shoulder Score (ASES score) | pretreatment, 24 weeks, 1 year, 2 year and 5 year
  Changes in patient self evaluation and physician assessment score
Veterans RAND Health (VR-12) | pretreatment, 24 weeks, 1 year, 2 year and 5 year
  Changes in patient reported general health and mental survey. Average score is 50 (negative answers bring scores down, positive answers bring score up)
Single Assessment Numerical Evaluation (SANE) | pretreatment, 24 weeks, 1 year, 2 year and 5 year
  Changes in patient reported affected shoulder survey base on percentage (0 - 100%, 100% being normal)
Visual Analogue Scale (VAS) | pretreatment, 24 weeks, 1 year, 2 year and 5 year
  Changes in patient reported pain survey. 0 - 10 point scale (0 no pain, 10 worst possible pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Southern Oregon Orthopedics, Medford, Oregon, United States

IPD SHARING:
Plan to Share IPD: No